CLINICAL TRIAL: NCT01904214
Title: A Single-dose, Open-label, Parallel-group Study to Assess the Pharmacokinetics of BAF312 in Subjects With Renal Impairment Compared to Subjects With Normal Renal Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CBAF312A2129
Record Dates: First submitted 2013-07-17; First posted 2013-07-22 (Estimated); Last update posted 2020-12-08 (Actual); Status verified 2018-02

CONDITIONS: Renal Impairment
Keywords: renal impairement; pharmacokinetics
MeSH Terms: conditions — Renal Insufficiency | interventions — siponimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- severe renal impairmnt (Experimental)
  Interventions: Drug: BAF312
- moderate renal impairment (Experimental)
  Interventions: Drug: BAF312
- mild renal impairment (Experimental)
  Interventions: Drug: BAF312
- healthy subjects (Experimental)
  Interventions: Drug: BAF312

INTERVENTIONS:
Drug: BAF312 — Treatment with a single oral dose of 0.25 mg BAF312

SUMMARY:
to quantify the effect of different degrees of renal impairment on the pharmacokinetics of BAF312 (and selected metabolites) and to assess safety and tolerability in order to develop dosing recommendations for subjects with renal impairment

ELIGIBILITY:
Inclusion Criteria:

All subjects:

* At least 50 kg and body mass index (BMI) within 18-38 kg/m2.
* CYP2C9 wild-type (CYP2C9*1 homozygous carriers)

Renal impairment:

- Subjects must have either mild, moderate or severe renal impairment

Exclusion Criteria:

All subjects

* Use of other investigational drugs within certain timelines
* Donation or loss of 400 mL or more of blood or plasma within eight (8) weeks prior to initial dosing
* History of cardiac rhythm abnormalities or cardiac rhythm abnormalities identified in the 24-h Holter ECG recording including episodes of bradycardia (HR < 50 bpm) during waking hours and/or arrhythmic episodes; subjects with history or presence of ventricular rhythm disturbances (ventricular extra-systoles >100/24h, or higher grade), or supraventricular arrhythmias (other than occasional supraventricular ectopic beats with a maximum of 5 subsequent ectopic beats per event) or subjects with conduction disturbances (higher than AV-block grade 1) or bradycardia or tachycardia.
* Women of child-bearing potential
* History of malignancy of any organ system
* History or presence of symptomatic postural hypotension or syncope.
* Total WBC or lymphocyte counts which falls outside the 1.5-fold local laboratory normal range or platelet count < 30,000/μL at screening or baseline.
* Clinically significant infection or recent vaccination with live-attenuated vaccines.
* History or presence of hepatitis B or C and/or positive Hepatitis B surface antigen (HBsAg) or Hepatitis C test result at screening.

Renal impairment:

* History or presence of any non-controlled and clinically significant disease that could affect the study outcome or that would place the patient at undue risk.
* Any surgical or medical condition other than renal impairment which might significantly alter the absorption, distribution, metabolism, or excretion of drugs, or which may jeopardize the safety of the study subject in case of participation in the study.
* Treatment with certain drugs

Healthy subjects:

* History or presence of any clinically significant disease of any major system organ class including (but not limited to) cardiovascular, metabolic, renal, neurological or psychiatric diseases.
* Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism, or excretion of drugs, drugs, or which may jeopardize the subject in case of participation in the study.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-07; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters of BAF312 and selected metabolites | pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72, 96, 144, 216, and 312 hours post dose
  The pharmacokineticsof BAF312 will be studied in plasma up to 312 (+/-24) hours post-dose at the following time points: pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72, 96, 144, 216, and 312 (+/-24) hours post dose. Selected metabolites will also be quantified using the same samples as described above. Free plasma circulating fraction of BAF312 will also be investigated to assess whether protein binding is affected by renal impairment. For this purpose a separate blood sample will be taken at the following time point: 4 hours post-dose.

SECONDARY OUTCOMES:
Number of participants with Adverse Events as a measure of Safety and Tolerability | Day 1 - Day 14
  Physical examination, vital signs, body temperature, standard safety laboratory evaluations (hematology, clinical chemistry, coagulation, Hepatitis B and C and HIV serology, pregnancy test, alcohol and drug screen), standard 12-lead electrocardiogram , cardiac monitoring, 24-h Holter ECG, (serious) adverse event monitoring.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- Novartis Investigative Site, Orlando, Florida, United States
- Novartis Investigative Site, Bucharest, Romania

REFERENCES:
- See also: Results for CBAF312A2129 can be found on the Novartis Clinical Trial Results website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=14230
- See also: Pubmed publication — https://www.ncbi.nlm.nih.gov/pubmed/27841151